CLINICAL TRIAL: NCT02080988
Title: Cross Sectional Evaluation of Coughing Force in Stroke Patients With Severe Aspiration
Brief Title: Reflexive Coughing Force in Severe Aspirators
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Sun Im, Assistant Professor, The Catholic University of Korea
Other Study IDs: HC 13OISE0066_2; BCMC13AH06 (Other: Bucheon St Mary's Hospital)
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Stroke
Keywords: stroke; deglutition disorders; cough; aspiration pneumonia; diaphragm; respiratory function
MeSH Terms: conditions — Stroke; Deglutition Disorders; Cough; Pneumonia, Aspiration; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Silent aspirators: Stroke patients with dysphagia with severe aspiration
- Non aspirating, no dysphagia group: Stroke patients with no dysphagia and no evidence of aspiration

SUMMARY:
To assess coughing force during reflex coughing test in those with severe dysphagia and severe aspiration and compare them to than those with stroke patients with no signs of dysphagia/aspiration.

DETAILED DESCRIPTION:
Severe aspiration with a compromised cough function can be a risk factor of aspiration pneumonia.

Reflexive coughing can be tested by administration of citric acid via a nebulizer. The objective of this study is to measure the cough force produced via citric acid inhalation challenge, and determine if those with severe aspiration with severe dysphagia have more weak cough force during reflexive cough testing that those post-stroke patients with no signs of aspiration or dysphagia after stroke.

We also aimed to measure the strenght of the respiratory measures with the use of surface EMG.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed stroke lesions
* Confirmed aspiration during vfss or fees examinations

Exclusion Criteria:

* Episode of acute pneumonia or pulmonary embolism at time of enrollment
* Previous history of chronic respiratory disorders or other systemic disorders that may affect respiratory function ( ex, rheumatoid disease, spinal cord injury)
* Stroke patients with multiple brain lesions
* Episode of Diaphragm weakness due to peripheral polyneuropathy or unilateral phrenic nerve palsy
* Previous episode of abdominal or thoracic surgery within one year of enrollment
* Concomitant diagnosis of myopathy, muscular dystrophy or other disorders that may affect respiratory muscles.
* Episode of rib fracture within one year of enrollment
* Chronic alcoholism
* Patient with previous diagnosis of dementia or with impaired cognitive function that may limit full participation at the evaluation
* Patient with tracheostomy state

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients with dysphagia with aspiration
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Coughing force | baseline one time
  Coughing force as assessed by reflexive cough test

SECONDARY OUTCOMES:
Coughing force during voluntary coughing | baseline one time

OTHER OUTCOMES:
Spirometry findings (Forced vital capacity, forced expiratory volume at one second) | baseline one time
Maximal inspiratory and expiratory pressure | baseline one time
Root mean square values of respiratory muscles | baseline one time
Diaphragm excursion as assessed by M mode sonography | baseline one time

CONTACTS AND LOCATIONS:
Overall Officials: Sun Im, Md PhD, Principal Investigator — The Catholic University of Korea; Geun Young Park, MD PhD, Study Chair — The Catholic University of Korea
Locations (1):
- Bucheon St Mary's Hospital, Bucheon-si, South Korea

REFERENCES:
- [Derived] Choi YM, Park GY, Yoo Y, Sohn D, Jang Y, Im S. Reduced Diaphragm Excursion During Reflexive Citric Acid Cough Test in Subjects With Subacute Stroke. Respir Care. 2017 Dec;62(12):1571-1581. doi: 10.4187/respcare.05488. Epub 2017 Sep 12. PMID 28900040